CLINICAL TRIAL: NCT04227431
Title: The Effect of Tresiba® (Insulin Degludec) in Type 2 Diabetes Patients in Real World Clinical Practice in China - Noninterventional, Retrospective Chart Review Study
Brief Title: A Research Study, Looking at How Tresiba® Works in People With Type 2 Diabetes in Local Clinical Practice in China
Acronym: CN-TREAT
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1250-4442; U1111-1208-5180 (Other: World Health Organization (WHO))
Record Dates: First submitted 2020-01-10; First posted 2020-01-13 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tresiba®: A broad real world type 2 diabetes (T2D) patient population in China, treated with oral anti-diabetic drugs (OAD(s)) or basal insulin prior to treatment initiation with Tresiba®
  Interventions: Other: Insulin degludec

INTERVENTIONS:
Other: Insulin degludec — Participants have been treated with Tresiba® (insulin degludec) for at least 20 weeks before entering the study. The study will be based on data already recorded in participants' medical records for approximately the last year and no new tests or procedures are required as part of the study.

SUMMARY:
The purpose of the study is to collect information on how Tresiba® works in patients with type 2 diabetes in China. The study will be based on data already recorded in participants' medical records and no new tests or procedures are required as part of the study. This study does not affect participants' current diabetes treatment. The study will look at data recorded in participants' medical records for approximately the last year. After signing the informed consent form, no further activities will be required from the participants.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent Form (ICF) obtained before any study-related activities. Study related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
* Male or female, aged at least 18 years at the time of signing the ICF.
* Diagnosed with T2D.
* Treated with any OAD(s) or basal insulin ± OAD(s), with or without prandial insulin for at least 20 weeks prior to treatment initiation with Tresiba®.
* The decision to initiate treatment with commercially available Tresiba® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.
* Treated with Tresiba® (with or without OADs, with or without prandial insulin) for at least 20 weeks and have at least one documented medical visit with HbA1c measurement in the first 20 weeks (plus/minus 8 weeks) after Tresiba® initiation. The patient may or may not be treated with Tresiba® at the time of patient selection to this study.
* Minimum available data: age, weight, and sex at the time of Tresiba® initiation, HbA1c (most recent value within 12 weeks prior to Tresiba® initiation and a value in the first 20 weeks [plus/minus 8 weeks] after Tresiba® treatment), and duration and type of insulin treatment (for insulin treated patients).

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having signed the ICF.
* Participation (defined as randomisation) in a diabetes clinical trial of an approved or non-approved investigational medicinal product within 20 weeks prior to the treatment initiation with Tresiba® or during the first 28 weeks of treatment with Tresiba®.
* Tresiba® not used in accordance with the local label.
* Patients treated with continuous subcutaneous insulin infusion or premix insulin in the 20 weeks prior to receiving Tresiba® (short-term [equal to or less than 14 days] treatment with continuous subcutaneous insulin infusion or premix insulin in the 20 weeks prior to receiving Tresiba® is allowed).
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetes Mellitus, Type 2 (T2D) patients, who had Tresiba® added to their previous Oral Anti-diabetic drugs (OADs) or were switched to Tresiba® treatment from any previous basal insulin based on the clinical judgement of the treating physician and were treated with Tresiba® for at least 20 weeks in routine clinical practice in China.
Sampling Method: Non-Probability Sample
Enrollment: 938 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2021-07-17 (Actual); Study Completion 2021-07-17 (Actual)

PRIMARY OUTCOMES:
Change in glycosylated haemoglobin (HbA1c) | Week 0, week 20
  Percent point

SECONDARY OUTCOMES:
Change in laboratory-measured fasting plasma glucose (FPG) | From baseline (week 0) to end of study (week 20)
  mmol/L
Change in self-measured fasting plasma glucose (SMPG) | From baseline (week 0) to end of study (week 20)
  mmol/L
Change in daily insulin doses (total, basal, prandial) | From baseline (week 0) to end of study (week 20)
  Units/day
Change in rates of hypoglycaemic episodes (number of episodes/patient years) (overall, nonsevere, severe, nocturnal) before and after add on of/switch to Tresiba® | From baseline (week 0) to end of study (week 20)
  Count. All recorded events will be captured in the 20 weeks prior to treatment initiation with Tresiba (week 0) and 20 weeks after treatments initiation with Tresiba (week 20)
Patient having at least one hypoglycaemic episode (overall, non-severe, severe, nocturnal) before and after add-on of/switch to Tresiba® (Yes/no) | From baseline (week 0) to end of study (week 20)
  Count
Change in number of concomitant non-insulin anti-diabetic drugs before and after add-on/switch to Tresiba® | From baseline (week 0) to end of study (week 20)
  Count. All recorded recorded concomitant non-insulin antidiabetic drugs will be captured in the 20 weeks prior to treatment initiation with Tresiba (week 0) and 20 weeks after treatments initiation with Tresiba (week 20)
Reason(s) for starting Tresiba®, at time of switch/add-on, if available | At baseline (week 20)
  Free text listing

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (56):
- China (56):
  - NIS-The Second Hospital of Anhui Medical Hospital, Hefei, Anhui
  - NIS-No.9 People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - NIS-The Third Affiliated Hospital of Chongqing Medical Univ., Chongqing, Chongqing Municipality
  - NIS-People's Hospital of Gansu Province, Lanzhou, Gansu
  - NIS-People's Hospital of Linxia, Gansu, Linxia, Gansu
  - NIS-Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - NIS-The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - NIS-Huizhou Third People's Hospital, Huizhou, Guangdong
  - NIS-Qingyuan People's Hospital, Qingyuan, Guangdong
  - NIS-Shenzhen Futian District People's Hospital, Shenzhen, Guangdong
  - NIS-The University of Hong Kong-Shenzhen Hospital, Shenzhen, Guangdong
  - NIS-General Hospital of Shenzhen University, Shenzhen, Guangdong
  - NIS-Hainan Provincial Hospital of TCM, Haikou, Hainan
  - NIS-People's Hospital of Henan Province, Zhengzhou, Hainan
  - NIS-Cangzhou Central Hospital, Cangzhou, Hebei
  - NIS-Dingzhou People's Hospital, Dingzhou, Hebei
  - NIS-CNPC Central Hospital, Langfang, Hebei
  - NIS-Langfang people's Hospital, Langfang, Hebei
  - NIS-The 3rd Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - NIS-Haerbin 1st Hospital, Harbin, Heilongjiang
  - NIS-The Second Affiliated Hospital of Harbin Medical Univ., Harbin, Heilongjiang
  - NIS-Heilongjiang Provincial Hospital, Harbin, Heilongjiang
  - NIS-The First Affiliated Hospital, Zhengzhou University, Zhengzhou, Henan
  - NIS-General Hospital of Shiyan Dongfeng Group, Shiyan, Hubei
  - NIS-Changzhou No.2 People's Hospital, Changzhou, Jiangsu
  - NIS-Kunshan 1st People's Hospital, Kunshan, Jiangsu
  - NIS-Nanjing Jiangbei Hospital, Nanjing, Jiangsu
  - NIS-The Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu
  - NIS-Zhong Da Hospital Southeast University, Nanjing, Jiangsu
  - NIS-Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - NIS-The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - NIS-Zhangjiagang Hospital of Traditional Chinese Medicine, Suzhou, Jiangsu
  - NIS-Wuxi 2nd People's Hospital, Wuxi, Jiangsu
  - NIS-No.2 Hospital Affiliated to Jilin University, Changchun, Jilin
  - NIS-The 1st Affi. Hosp. of Changchun Univer. of Chinese Medi, Changchun, Jilin
  - NIS-People's Hospital of Liaoning Province, Shenyang, Liaoning
  - NIS-Shenyang Central Hospital, Shenyang, Liaoning
  - NIS-The Affiliated Hospital of Liaoning TCM University, Shenyang, Liaoning
  - NIS-The 4th Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - NIS- Qinghai Red Cross Hospital, Xining, Qinghai
  - NIS-Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shaanxi
  - NIS-Second Hospital of Shanxi Medical University, Taiyuan, Shaanxi
  - NIS-Affiliated Hospital of Shanxi TCM Colleage, Xianyang, Shaanxi
  - NIS-Affiliated Hospital of Shanxi Yanan Medical Colleage, Yan’an, Shaanxi
  - NIS-Weifang People's Hospital, Weifang, Shandong
  - NIS-Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - NIS-No.1 Hospital affiliated to Shihezi Medical College, Shihezi, Xinjiang
  - NIS-Xinjiang Traditional Chinese Medicine Hospital, Ürümqi, Xinjiang
  - NIS-The 5th Affiliated Hospital of Xinjiang Medical Univ., Ürümqi, Xinjiang
  - NIS-The 2nd Affiliated Hospital of Xinjiang Medical Univer., Ürümqi, Xinjiang
  - NIS-The First Affiliated Hospital of Xinjiang Medical Univ., Ürümqi, Xinjiang
  - NIS-Dali First People's Hospital, Dali, Yunnan
  - NIS-The Second Affiliated Hospital of Kunming Medical Univ., Kunming, Yunnan
  - NIS-Ningbo First Hospital, Ningbo, Zhejiang
  - NIS-The No.2 Hospital affiliated to Guizhou Medical college, Kaili
  - NIS-People's Hospital of Qinghai Province, Xining

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Wang W, Chang X, Lehrskov LL, Li L, Nordentoft M, Quan J, Sha Y, Zhong X, Yang C, Zhu D. Insulin Degludec in People with Type 2 Diabetes in China: A Non-interventional, Retrospective Chart Review Study (CN-TREAT). Diabetes Ther. 2024 Mar;15(3):725-739. doi: 10.1007/s13300-024-01533-6. Epub 2024 Mar 5. PMID 38438707